CLINICAL TRIAL: NCT04061109
Title: Multicenter, Noncontrol Study of Recombinant Coagulation Factor VIII for Prophylactic Therapy in Subjects With Hemophilia A.
Brief Title: Safety, Efficacy Evaluation of Recombinant Coagulation Factor VIII Injection in Subjects With Hemophilia A.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CTTQ-NXBYZ-02
Record Dates: First submitted 2019-07-16; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prophylactic therapy (Experimental): Subjects received Recombinant Human Coagulation FVIII for prophylactic therapy with 25 - 35 IU/kg injection once every other day or three times per week for 6 months.
  Interventions: Drug: Recombinant Human Coagulation FVIII

INTERVENTIONS:
Drug: Recombinant Human Coagulation FVIII — A kind of Recombinant Coagulation Factor VIII Injection produced by sponsor.

SUMMARY:
This is a multi-center, open-label, single-arm trial to evaluate the efficacy and safety of Recombinant Coagulation Factor VIII in patients with hemophilia A . Recombinant Coagulation Factor VIII is prophylactic administrated 25 - 35 IU/kg once every other day or three times per week which should be continuous for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Hemophilia A.
2. FVIII:C <1%. 3）12 and 65 years old.

4）Has received FVIII treatment and the treatment exposure days ≥100. 5）Has bleeding treatment records of at least 3 months before randomization. 6）FVIII inhibitor assay results is negative. 7） Subjects should agree to use an adequate method of contraception during the study.

8）Understood and Signed an informed consent form.

Exclusion Criteria:

1. Has a history or family history of blood coagulation factor VIII inhibitor.
2. Has other coagulation dysfunction diseases in addition to hemophilia A.
3. HIV positive.
4. Plan to receive surgery during the trial.
5. Has used immunomodulator within one weeks before the first dose，and less than 7 half-life periods.
6. Known to be allergic to experimental drugs or any excipients.
7. Severe anemia and need blood transfusion.
8. Serious liver or kidney damage.
9. Serious heart disease.
10. Uncontrollable hypertension.
11. Has participated in other clinical studies within one month before the first dose.
12. The researchers believe that it is not suitable for participants.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Annualized joint bleeding rate | up to 24 weeks
  Annualized joint bleeding rate（AJBR） can be calculated using the following formula: Number of joint bleeding events during efficacy evaluation period/(number of days in treatment period/365.25).
Incremental Recovery of the First Dose | After the first dose on day 1
  Peak activity of FVIII (as Cmax) measured within 1 hour after the end of injection

SECONDARY OUTCOMES:
Bleeding Event Treatment Efficacy | up to 24 weeks
  The investigator shall evaluate the hemostatic effect after the treatment of every bleeding event of subjects based on a four-point scale(excellent, good, moderate, not relieved).
Monthly Average Number of Bleedings | up to 24 weeks
  Number of bleeding events in each month.
The number and dose of injection of Recombinant Human Coagulation FVIII required per bleeding episode | up to 24 weeks
  The number and dose of injection of Recombinant Human Coagulation FVIII required per bleeding episode
Incremental Recovery of Duplicated Dose | up to 12 weeks, 24 weeks
  Peak activity of FVIII (as Cmax) measured within 1 hour after the end of injection.
Hemophilia Joint Health Score (HJHS) | Baseline, week 24
  The scale assesses the functional status of the six major joints of the elbow, knee, and ankle, including: joint swelling, swelling duration, muscle atrophy, muscle strength, joint friction, joint pain, joint extension, joint flexion Degree decline, overall gait, etc.
Assess the impact of Recombinant Human Coagulation FVIII following Patient Reported Outcome (PRO) EQ-5D | Baseline, week 24
  EQ-5D is a general questionnaire designed to measure health status on a scale of 0-100 with the higher value representing a better outcome and record the participants' current health state in 5 domains mobility, selfcare, usual activities, pain, anxiety.

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - AnHui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - FuJian Medical University Union Hospital, Fuzhou, Fujian
  - The First Hospital of LanZhou University, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - HeNan Provincial Peoples Hospital, Zhengzhou, Henan
  - HeNan Cancer Provincial Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality